CLINICAL TRIAL: NCT05258812
Title: Cytopenias in Hospitalized Patients of COVID-19 During First and Other Waves
Brief Title: Cytopenias in Hospitalized Patients of Corona Virus Infection(COVID-19) During First and Other Waves
Status: Completed | Type: Observational
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ambreen Kashif, Doctor, Fatima Memorial Hospital
Other Study IDs: FMH
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Corona Virus Infection
Keywords: COVID-19; Cytopenia; Thrombocytopenia; Anemia; Leucopenia
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Cytopenia; Thrombocytopenia; Anemia; Leukopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Demographic, Clinical and laboratory data as well as outcome of total 202 COVID-19 patients who were Polymerase Chain Reaction (PCR) positive and admitted in Fatima memorial Hospital, Lahore, Pakistan, was collected during first and other waves. Data of First wave is from May 2020 to July 2020, second wave from early November to Mid December 2020 and third wave from Mid march to June 2021. Investigator analyzed the data on basis of Systemic immune inflammatory index (SII) as well hematological parameters of First Wave were compared to other waves of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 Positive Hospitalized patients
* All genders

Exclusion Criteria:

* Patients with Known hematological disorders
* Patients with known chronic Liver Disease

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 Positive Hospitalized patients, of all genders and all age group.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Cytopenias in Hospitalized Patients of COVID-19 During First and Other waves | 4 weeks
  extent of cytopenias is being measured in COVID-19 hospitalized patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima memorial Hospital, Lahore, Punjab Province, Pakistan

DOCUMENTS (1):
  • Study Protocol (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT05258812/Prot_000.pdf